CLINICAL TRIAL: NCT00637026
Title: A PreSurgical Study to Evaluate Molecular Alterations That Occur in Human Breast Cancer Tissue and Normal Skin After Short Term Exposure to ZD1839 (IRESSA) and to Correlate These Alterations With Pharmacokinetic Parameters.
Brief Title: Ph II Early BC Pre-Surgical Biologic Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Cancer International Research Group (CIRG) (Other)
Responsible Party: Alison Armour Medical Science Director, AstraZeneca
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1839IL/0219
Record Dates: First submitted 2008-03-10; First posted 2008-03-17 (Estimated); Last update posted 2009-04-23 (Estimated); Status verified 2009-04

CONDITIONS: Breast Cancer
Keywords: Iressa, Gefitinib, Breast Cancer, Surgery
MeSH Terms: conditions — Breast Neoplasms | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Gefitinib — Iressa

SUMMARY:
A pre-surgery study to assess changes that occur in human breast cancer material and normal skin after a short course of treatment with Iressa.

ELIGIBILITY:
Inclusion Criteria:

* Invasive breast cancer, Aged 18 years or older, Not more than 28 days from initial diagnosis

Exclusion Criteria:

* Pregnant or lactating patients, Prior or current radiotherapy for breast cancer, Known allergy reaction to Iressa

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2003-07; Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Molecular alterations occuring in breast cancer tissue following Iressa treatment | At time of diagnosis and time of patient surgery

SECONDARY OUTCOMES:
Molecular alterations occurring in normal skin tissue following Iressa treatment | At time of diagnosis and time of patient surgery
To correlate molecular changes with pharmacokinetic parameters | At time of diagnosis and time of patient surgery
To evaluate tolerability of short term Iressa treatment